CLINICAL TRIAL: NCT04907643
Title: Randomized Controlled Trial of Virtual Reality for GI Cancer Pain to Improve Patient Reported Outcomes
Brief Title: Virtual Reality for GI Cancer Pain to Improve Patient Reported Outcomes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Brennan Spiegel, Director of Health Services Research, Cedars-Sinai Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: STUDY00001363; R01CA252211 (NIH)
Record Dates: First submitted 2021-01-26; First posted 2021-06-01 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Cancer Pain; Visceral Pain; Gastrointestinal Neoplasms; Cancer of Gastrointestinal Tract; Small Intestine Cancer; Pancreas Cancer; Liver Cancer; Colon Cancer; Biliary Tract Cancer; Stomach Cancer; Rectum Cancer; Peritoneal Cancer; Gastrointestinal Cancer Metastatic; Gastrointestinal Cancers - Anus; Gastrointestinal Cancers - Stomach; Gastrointestinal Cancers - Colorectal; Gastrointestinal Cancers - Small Intestine; Small Intestine Cancer Stage III; Small Intestine Cancer Stage IV; Small Intestine Cancer, Recurrent; Pancreas Cancer, Stage III; Pancreas Cancer, Stage IV; Pancreas Cancer, Metastatic; Pancreas Cancer, Recurrent; Liver Cancer Stage IIIa; Liver Cancer Stage IIIb; Liver Cancer Stage IIIc; Liver Cancer Stage IV; Colon Cancer Stage III; Colon Cancer Stage IV; Stomach Cancer Stage III; Stomach Cancer Stage IV; Stomach Cancer Recurrent; Rectum Cancer, Recurrent; Gastrointestinal Cancers - Liver; Anal Cancer; Anal Cancer Stage III; Anal Cancer Stage IV; Anal Cancer Recurrent; Anal Cancer Metastatic; Anal Cancer, Stage IIIA; Anal Cancer, Stage IIIB; Appendix Cancer; Ampullary Cancer; Bile Duct Cancer; Bile Duct Cancer Stage III; Bile Duct Cancer Stage IV; Bile Duct Cancer Stage IVA; Bile Duct Cancer Stage IVB; Bile Duct Cancer Recurrent; Carcinoid Tumor; Carcinoid Tumor of Pancreas; Carcinoid Tumor of Large Intestine; Carcinoid Tumor of GI System; Carcinoid Tumor of Colon; Carcinoid Tumor of Liver; Carcinoid Tumor of Cecum; Carcinoid Tumor of Ileum; Carcinoid Tumor of Rectum; Carcinoid Tumor of the Small Bowel; Carcinoid Tumor of the Stomach; Large Intestine Cancer; Esophagus Cancer; Esophagus Cancer, Stage III; Esophagus Cancer, Stage IV; Esophagus Cancer, Recurrent; Gallbladder Cancer; Gallbladder Cancer Stage III; Gallbladder Cancer Stage IV; Gastric (Stomach) Cancer; Neuroendocrine Tumor; Peritoneum Cancer; Rectal Cancer; Esophagus Cancer, Stage I; Esophagus Cancer, Stage II; Gallbladder Cancer Stage I; Gallbladder Cancer Stage II; Bile Duct Cancer Stage I; Bile Duct Cancer Stage II
Keywords: Virtual Reality; VR; support; GI cancer; cancer pain
MeSH Terms: conditions — Cancer Pain; Visceral Pain; Gastrointestinal Neoplasms; Pancreatic Neoplasms; Liver Neoplasms; Colonic Neoplasms; Biliary Tract Neoplasms; Stomach Neoplasms; Rectal Neoplasms; Recurrence; Neoplasm Metastasis; Anus Neoplasms; Appendiceal Neoplasms; Bile Duct Neoplasms; Carcinoid Tumor; Esophageal Neoplasms; Gallbladder Neoplasms; Neuroendocrine Tumors

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (3):
- Virtual Reality Program A (Experimental): This arm will include software that provides immersive skills-based content for pain reduction.
  Interventions: Device: PICO G2 4k
- Virtual Reality Program B (Experimental): This arm will include software that provides immersive distraction based content for pain reduction.
  Interventions: Device: PICO G2 4k
- Virtual Reality Program C (Sham Comparator): This arm will include software that provides nonimmersive distraction based content for pain reduction.
  Interventions: Device: PICO G2 4k

INTERVENTIONS:
Device: PICO G2 4k — Participants will use the Pico G2 4K VR audio and visual head-mounted device. The Pico G2 4K is a standalone VR headset that comes with an orientation-tracked controller. It does not require a smartphone or personal computer to operate. The device supports 3 degrees of freedom (3DOF) head tracking, has best-in-class optics, and a wide field-of-view.

SUMMARY:
Patients with digestive tract malignancy often experience severe and unremitting abdominal pain that negatively affects physical, emotional, and social function, as well as health related quality of life (HRQOL). Therapeutic virtual reality (VR) has emerged as a promising and evidence-based treatment modality for cancer pain. Users of VR wear a pair of goggles with a close-proximity screen in front of the eyes that creates a sensation of being transported into lifelike, three-dimensional worlds. To date, VR has been limited to short-term clinical trials for cancer pain. Moreover, limited research exists on theory-based VR modalities beyond mere distraction, such as VR that employs acceptance and commitment therapy (ACT) with components of biofeedback and mindfulness. To bridge these gaps, this study seeks to: (1) assess the impact of immersive VR on patient-reported outcomes (PROs), including pain, activity metrics, and opioid use among patients with visceral pain from a digestive tract malignancy; (2) assess differences in PROs, activity metrics, and opioid use between skills-based VR therapy vs. distraction VR therapy; and (3) determine patient-level predictors of VR treatment response in visceral cancer pain.

To address these aims, the study will measure PROs and opioid use in 360 patients randomized among 3 groups and follow them for 60 days after enrollment: (1) an enhanced VR group receiving skills-based VR; (2) a distraction-based VR group receiving patient-selected VR videos; and (3) a VR sham control group using a VR headset with 2-D content. The results will inform best practices for the implementation of VR for visceral cancer pain management and guide selection of patient-tailored experiences.

DETAILED DESCRIPTION:
GI cancer pain is a prevalent and costly condition. Medical therapy is not always effective for managing GI cancer pain; there is a need for drug-free alternative to complement or even replace medical therapy, such as opioids. This study will evaluate a novel technology called virtual reality (VR). Users of VR wear a pair of goggles with a three-dimensional screen that creates a sensation of being transported into lifelike worlds. Evidence shows that VR can reduce pain through many different mechanisms. Research shows that VR can also help train people in new skills, such as to meditate, breathe deeply, and learn how to cope with pain.

In this study, patients with GI cancer pain will be randomized into three groups of equal size: (1) immersive skills-based VR therapy; (2) immersive distraction VR therapy; and (3) non-immersive sham VR using 2D videos displayed in a VR headset. The skills-based treatment will use virtual healing environments to teach patients about meditation, breathing exercises, and pain management. The distraction treatment will use immersive videos that are designed to take the mind off of pain. The sham VR will use VR goggles, but patients will only watch a two-dimensional video rather than a 3D, immersive experience.

Eligible patients will have GI cancer pain, meaning belly pain at least 5 points above the national average on the NIH PROMIS GI Scale as well as having a GI cancer diagnosis. . The study will exclude people who are under 18 years of age, unable to understand the consent form, expected to live less than 3 months, brain tumors not responding to treatment, or injury that makes it difficult to wear something on their face.

Randomization between groups will occur using a computer program called REDCap and will be performed after obtaining patient consent for participating in the study. The VR goggles will be shipped via FedEx to patients in all three groups, along with instructions for use. Patients will then be asked to actively use the headset for four weeks on a daily basis, following the specific instructions for their assigned intervention. In addition, patients will wear a Fitbit watch on their wrist during the study, as tolerated, to monitor step counts and sleep. Participants will fill out a set of weekly questionnaires that will be sent via email.

In order to show a difference between the active VR treatments and the sham VR control treatment, the investigator will recruit a minimum of 120 patients in each arm of the study. This calculation is sufficient to demonstrate clinically meaningful differences in the primary outcome, which is Gastrointestinal belly pain levels as measured by the NIH Patient Reported Outcome Measurement Information System, or PROMIS® questionnaire. PROMIS is a well-validated set of questionnaires that measure different aspects of quality of life; for this study the investigator will focus on PROMIS Gastrointestinal belly pain, Global physical and mental health, and Social isolation. Daily pain catastrophizing, Milligram morphine equivalent daily dose, Simulator sickness, Pain treatment satisfaction, Pain self-efficacy (PSEQ), baseline demographic information, Pain Diary, and Pain Behaviors will also be measured. The investigator will compare the number of steps taken per day and sleep levels among the three groups using statistical tests that account for potential difference among the groups. Finally, the investigator will perform statistical analyses to identify whether there are individual patient characteristics that predict response to VR therapy. The goal will be to develop a mathematical algorithm that optimized patient selection to make more precise treatment decisions with VR.

To learn more about the study and to assess your eligibility, please visit our study website at: https://virtualmedicine.org/research/current/gicancer

ELIGIBILITY:
Inclusion Criteria:

* Have a primary malignancy of the biliary tract, colon, liver, pancreas, peritoneum, rectum, small intestine, or stomach, with no plan for resection during the study period
* Tumor types including, but not limited to, adenocarcinoma, squamous cell carcinoma, neuroendocrine tumors, and tumors of mesenchymal origin will be eligible
* Have clinically significant visceral pain, measured using the standardized NIH PROMIS GI Pain Scale defined as scoring at least 5 points above the nationally normed score
* Ability to read and write in English

Exclusion Criteria:

* Have a condition that interferes with VR usage, including but not limited to seizures, facial injury precluding safe placement of headset, and visual impairments
* Have cognitive impairment that affects protocol participation. This will be done with a three part cognitive assessment during the initial phone call to assess eligibility followed by consent discussion if eligible.
* Have brain metastases
* Have a prognosis of <3 months from the time of enrollment per treating oncologist

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2021-10-05 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-06-16 (Estimated)

PRIMARY OUTCOMES:
Patient-Reported Outcomes Measurement Information System Gastrointestinal Belly Pain over 30 days from the baseline | Over 30 days from the baseline
  Gastrointestinal Belly Pain over time as measured by Patient-Reported Outcomes Measurement Information System Gastrointestinal Belly Pain 5a delivered on a weekly basis (T-Scored, Continuous, 1-5, higher the worse).

SECONDARY OUTCOMES:
Patient-Reported Outcomes Measurement Information System Gastrointestinal Belly Pain | Over 60 days
  Gastrointestinal Belly Pain over time as measured by Patient-Reported Outcomes Measurement Information System Gastrointestinal Belly Pain 5a delivered on a weekly basis (T-Scored, Continuous, 1-5, higher the worse).
Daily pain intensity | At baseline, week of Day 30, and week of Day 60
  Daily pain intensity for one week at baseline, week of Day 30, and week of Day 60 as measured by Daily Pain Intensity Scale (0-10, where 0 means no pain and 10 means the worst pain imaginable).
Patient-Reported Outcomes Measurement Information System Global physical and mental health | Over 60 days
  Global physical and mental health over time as measured by Patient-Reported Outcomes Measurement Information System Global Physical and Mental 2a. delivered on a weekly basis (1-5, higher the better)
Opioid prescriptions of Morphine Milligram Equivalents (MME) | In a 60-day period
  Comparing the change from study baseline to Day 60 in weekly MME of prescribed medication.

OTHER OUTCOMES:
Patient-Reported Outcomes Measurement Information System Pain Interference 4a | Over 60 days
  Pain interference over time as measured by Patient-Reported Outcomes Measurement Information System-Pain Interference 4a delivered on a weekly basis (T-Scored, Continuous, 1-5, higher the worse).
Patient Global Impression of Change | Over 60 days
  Patient Global Impression of Change over time as measured by Patient Global Impression of Change Scale delivered on a weekly basis (PGIC, 1-7, higher the worse).
Patient-Reported Outcomes Measurement Information System Social Isolation | Over 60 days
  Social Isolation over time as measured weekly by Patient-Reported Outcomes Measurement Information System Social Isolation short form 4a. delivered on a weekly basis (1-5, higher the worse)
Pain Catastrophizing scale 4 item short form. | Over 60 days
  Pain catastrophizing over time as measured by Pain Catastrophizing scale (PCS) 4 item short form delivered on a weekly basis (0-4, from not at all to all the time, higher the worse).
Steps taken per day | Continuous for 60 days
  Steps taken per day over time as measured by Fitbit smartwatch.
Minutes of sleep over time | Continuous for 60 days
  Minutes of sleep over time as measured by Fitbit smartwatch.
Pain coping skills survey | Day 60
  Assessment of pain coping skills over time as measured by a custom pain coping skills survey.
Pain Self-Efficacy Questionnaire (PSEQ) 2-item short form | Over 60 days
  Pain self-efficacy over time as measured by The Pain Self-Efficacy Questionnaire (PSEQ) 2-item short form delivered on a weekly basis (0-6, higher the better).
Dosage of VR (minutes per week) | Continuous for 60 days
  minutes of use per week will be extracted from the VR device via wifi network

CONTACTS AND LOCATIONS:
Overall Officials: Brennan Spiegel, MD, MSHS, Principal Investigator — Cedars-Sinai Medical Center; Scott Irwin, MD, PhD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- See also: Study web portal for more information and a self-assessment for eligibility — https://virtualmedicine.org/research/current/gicancer